CLINICAL TRIAL: NCT06767943
Title: Clinical Scoring and Biomarkers for Prediction of Myocardial Infarction After Non-Cardiac Surgery (MINS) Syndrome in Patients Undergoing Major Abdominal Surgeries
Brief Title: Predicting Myocardial Infarction After Abdominal Surgery: Clinical Scores & Biomarkers
Status: Completed | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Mohammed Abd ElRahman Hammed, Assistant Lecturer of Anesthesia, Pain & ICU, Benha University
Other Study IDs: Rc 6-11-2024
Record Dates: First submitted 2025-01-06; First posted 2025-01-10 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — Electrocardiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Myocardial Infarction After Non-Cardiac Surgery (MINS) Syndrome Group
  Interventions: Diagnostic Test: 12-lead electrocardiography

INTERVENTIONS:
Diagnostic Test: 12-lead electrocardiography — All patients were admitted to the intermediate care unit for the 1st 24-h PO for follow-up for the possibility of developing acute myocardial infarction (AMI), which was diagnosed according to the 2017 ESC Guidelines; by 12- lead electrocardiography

SUMMARY:
All patients undergoing non-cardiac surgery who met the inclusion criteria underwent a preoperative evaluation using specific assessment tools.

Following surgery, patients were closely monitored in the intermediate care unit for the first 24 hours for the development of acute myocardial infarction (AMI). AMI was diagnosed based on the presence of chest pain, elevated cardiac biomarkers, and specific electrocardiogram (ECG) and echocardiogram findings.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 45,
* Patients of ASA-PS grade II-IV,
* Patients who prepared for non-cardiac surgeries of SSS of II-IV,
* Patients free of exclusion criteria,
* Patients signed the written consent for the study precipitation.

Exclusion Criteria:

* Patients of ASA-PS grade I or V,
* Patients younger than 60 years,
* Patients planned to undergo surgeries of SSS >IV,
* Patients were severely frail with CFS>6,
* Patients had abnormal preoperative electrocardiography (ECG),
* Patients had a history of previous major cardiac or cerebrovascular events,
* Patient had disturbed cognitive function, coagulopathy, severe anemia with hemoglobin concentration (HBC) < 7 gm/dl.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients assigned for non-cardiac surgeries who fulfilled the inclusion criteria underwent preoperative evaluation using the assessment tools. All patients were admitted to the intermediate care unit for the 1st 24-h PO for follow-up for the possibility of developing acute myocardial infarction (AMI), which was diagnosed according to the 2017 ESC Guidelines and was differentiated as STEMI and NSTEMI.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
The proportion of patients reported having at least a 50% incidence of Myocardial Infarction (measured by the Relevant Changes in 12-Leads ECG) in correlation with blood biomarkers. | 50 Days
  The incidence of Myocardial infarction after major abdominal surgery detected by relevant changes in 12 leads ECG and in correlation to presence of blood biomarkers

CONTACTS AND LOCATIONS:
Locations (1):
- Benha University, Banhā, El Qalyoubia, Egypt